CLINICAL TRIAL: NCT01124929
Title: A Multi-centric Study on Treatment of Abdominal Tuberculosis (Intestinal or Peritoneal): A Randomized Controlled Trial to Compare the 6 Months of Cat I Treatment With 9 Months of Cat I Treatment (Extension for 3 Months) in Abdominal Tuberculosis Under the Revised National Tuberculosis Control Program
Brief Title: Treatment Duration for Abdominal Tuberculosis
Acronym: RNTCP-DOTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government); Christian Medical College, Vellore, India (Other)
Responsible Party: Principal Investigator, Govind K Makharia, Additional Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Abdominal TB_RCT (RNTCP-DOTS)
Record Dates: First submitted 2010-05-03; First posted 2010-05-18 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Tuberculosis
Keywords: Intestinal tuberculosis; Tuberculous peritonitis; Abdominal tuberculosis
MeSH Terms: conditions — Tuberculosis; Peritonitis, Tuberculous

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Category I treatment for 6 months (Active Comparator): Anti-tuberculosis drugs
  Interventions: Drug: RNTCP Category I treatment for 6 months
- Arm 2: Category I treatment for 9 months (Active Comparator): Anti-tuberculosis drugs,
  Interventions: Drug: RNTCP Category I treatment for 9months

INTERVENTIONS:
Drug: RNTCP Category I treatment for 6 months — 2H3R3Z3 E3 + 4H3R3
  Arms: Arm 1: Category I treatment for 6 months
Drug: RNTCP Category I treatment for 9months — 2H3R3Z3 E3 + 7H3R3
  Arms: Arm 2: Category I treatment for 9 months

SUMMARY:
Most of the guidelines on the treatment of tuberculosis suggest that 6 months treatment is sufficient for extrapulmonary tuberculosis except for bone tuberculosis and tubercular meningitis. Despite these recommendations, most physicians treating abdominal tuberculosis use antituberculous therapy for 9 months, sometimes even 12 months without any scientific justification. In a randomized controlled trial, Balasubramaniam et al reported no difference in success rate of 6mo (99%) vs 12 months (94%) antituberculous drugs (conventional strategy) in the treatment of abdominal tuberculosis.

Although Directly Observed Therapy (DOTs) have been proved to be effective in patients with pulmonary tuberculosis, lymph nodal tuberculosis, however, there is a lack of data on efficacy of DOTS in other extra-pulmonary disease including abdominal tuberculosis. Therefore, there is an urgent need to establish the efficacy of DOTs strategy of antituberculous therapy in the treatment of abdominal tuberculosis.

Therefore, the investigators planned to conduct a multicenter randomized controlled trial to determine the difference in the recurrence of disease after only observation for three months and three months extension of DOTs in a subset of patients with definite clinical response after 6 months of DOTs.

DETAILED DESCRIPTION:
Rationale Most of the guidelines on the treatment of tuberculosis suggest that 6 months treatment is sufficient for extrapulmonary tuberculosis except for bone tuberculosis and tubercular meningitis. Despite these recommendations, most physicians treating abdominal tuberculosis use antituberculous therapy for 9 months, sometimes even 12 months without any scientific justification. In a randomized controlled trial, Balasubramaniam et al reported no difference in success rate of 6mo (99%) vs 12 months (94%) antituberculous drugs (conventional strategy) in the treatment of abdominal tuberculosis.

Although DOTS have been proved to be effective in patients with pulmonary tuberculosis, lymph nodal tuberculosis, however, there is a lack of data on efficacy of DOTS in other extra-pulmonary disease including abdominal tuberculosis. The aim of the present study is not to assess the efficacy of DOTs but whether the Cat I regimen for 6 months is effective in the treatment of abdominal tuberculosis. We, therefore planned to conduct a multicenter randomized controlled trial to determine the difference in the efficacy and recurrence rate in 6months and 9 months of intermittent short course category I regimen under RNTCP.

Hypothesis There may not be a significant difference in the efficacy and recurrence rate of abdominal tuberculosis in those treated for six months vs those treated for 9 months with intermittent short course category I regimen under RNTCP.

Objectives

Primary objectives:

1. To determine the efficacy of intermittent short course chemotherapy for 6 months under Directly Observed Therapy (Category I under RNTCP) in treatment of abdominal tuberculosis (proportion of patients responding to treatment)
2. To determine difference in the recurrence of disease between the two randomized groups after only observation for three months and extension of RNTCP Cat I for three months in a subset of patients with definite clinical response after 6 months of DOTs Secondary objective

1. To study the effect of anti-tubercular drugs on the natural history of intestinal stricture due to tuberculosis Outcomes

Outcome measures:

Primary:

1. Response to treatment (6 months and nine months of RNTCP Cat I treatment) as defined earlier
2. Recurrence of symptoms of abdominal tuberculosis (intestinal and peritoneal) after 1 year of follow up in those who receive 6 months or 9 months of Cat I treatment.

ELIGIBILITY:
Inclusion criteria:

* Newly diagnosed patients with Intestinal TB or Peritoneal TB
* Has not received ATT for Tuberculosis any where in the body during past 5 years
* Patients having good general health and not too sick.
* Patients willing and likely to comply with the study procedures and follow up
* Patients should give informed consent.

Exclusion Criteria:

* Eighteen year is a cut off age for definition of adult and pediatric and adolescent medicine. The dosing of drugs are different in these two age groups. Therefore we plan to include patients of more than 18 years of age with abdominal TB in this study.
* Intake of ATT during the past 5 years
* Doubtful diagnosis
* Crohn's disease
* Patients with HIV and AIDS may have another systemic opportunistic infections including GI infections like cryptosporidiosis, Microsporidiosis or isosporiasis. There may be an overlap of GI manifestations such as diarrhea, abdominal pain, anemia, fever. Therefore, assessment of response to anti-tuberculosis therapy may be blurred. In order to keep the study group homogenous for comparison, we plan to exclude all those with HIV infection
* Chronic Liver Disease
* Associated significant co-morbidities
* H/O Sensitivity
* Peritoneal carcinomatosis
* Patients must not been used investigational agents during the past 6 months
* Unwilling patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Response to treatment (after 6 months and nine months of RNTCP Category I treatment) | 1 year
  Intestinal tuberculosis:
  Complete response to treatment: Resolution of clinical manifestations, Healing of demonstrable lesions, Microbiological response (Conversion of positive to negative)
  Clinical failure: Failure of response to treatment:
  Persistence of clinical manifestations Persistence of morphological lesions
  Peritoneal tuberculosis: Definition for response Complete response: Complete resolution of ascites within 6 months No response: Persistence of ascites
Recurrence of symptoms of abdominal tuberculosis (intestinal and peritoneal) after 1 year of follow up in those who receive 6 months or 9 months of Cat I treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr Govind K Makharia, MD, DM, DNB, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Dr Govind K Makharia, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Makharia GK, Ghoshal UC, Ramakrishna BS, Agnihotri A, Ahuja V, Chowdhury SD, Gupta SD, Mechenro J, Mishra A, Mishra A, Pathak MK, Pandey RM, Sharma R, Sharma SK. Intermittent Directly Observed Therapy for Abdominal Tuberculosis: A Multicenter Randomized Controlled Trial Comparing 6 Months Versus 9 Months of Therapy. Clin Infect Dis. 2015 Sep 1;61(5):750-7. doi: 10.1093/cid/civ376. Epub 2015 May 12. PMID 25969531